CLINICAL TRIAL: NCT04488419
Title: A Randomized, Placebo-Controlled, Double-Blind Study of ATH-1017 Treatment in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: ATH-1017 for Treatment of Mild to Moderate Alzheimer's Disease
Acronym: LIFT-AD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Athira Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATH-1017-AD-0201
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Dementia of Alzheimer Type
Keywords: Alzheimer's Disease; Cognition; Dementia; ATH-1017; LIFT AD; Fosgonimeton
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dosage (Experimental): Daily subcutaneous (SC) injection of 40mg ATH-1017
  Interventions: Drug: ATH-1017
- Placebo (Placebo Comparator): Daily subcutaneous (SC) injection of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATH-1017 — Daily subcutaneous (SC) injection of ATH-1017 in a pre-filled syringe
  Arms: Dosage
Drug: Placebo — Daily subcutaneous (SC) injection of Placebo in a pre-filled syringe
  Arms: Placebo

SUMMARY:
This study is designed to evaluate safety and efficacy of fosgonimeton (ATH-1017) in the treatment of mild to moderate Alzheimer's disease with a randomized treatment duration of 26-weeks.

DETAILED DESCRIPTION:
The study is designed to evaluate safety and efficacy of ATH-1017 in mild to moderate AD subjects, with randomized, parallel-arm treatment duration of 26 weeks, and based on clinical diagnostic criteria of Alzheimer's disease. Clinical efficacy is demonstrated by improvement in cognition and global/functional assessments comparing treatment to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 55 to 85 years
* Mild-to-moderate AD dementia subjects, MMSE 14-24, CDR 1 or 2 at Screening
* Clinical diagnosis of dementia, due probably to AD, by Revised National Institute on Aging-Alzheimer's Association criteria (McKhann, 2011)
* Body mass index (BMI) of ≥ 18 and ≤ 35 kg/m2 at Screening
* Reliable and capable support person/caregiver
* Treatment-free (subjects not receiving acetylcholinesterase inhibitor [AChEI] treatment), defined as:

  * Treatment-naïve, OR
  * Subjects who received an AChEI in the past and discontinued at least 4 weeks prior to Screening

Key Exclusion Criteria:

* History of significant neurologic disease, other than AD, that may affect cognition, or concurrent with the onset of dementia
* Subject has atypical variant presentation of AD, if known from medical history, particularly non-amnestic AD
* History of brain MRI scan indicative of any other significant abnormality
* Diagnosis of severe major depressive disorder even without psychotic features.
* Significant suicide risk
* History within 2 years of Screening, or current diagnosis of psychosis
* Myocardial infarction or unstable angina within the last 6 months
* Clinically significant cardiac arrhythmia (including atrial fibrillation), cardiomyopathy, or cardiac conduction defect (note: pacemaker is acceptable)
* Subject has either hypertension or symptomatic hypotension
* Clinically significant ECG abnormality at Screening
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) <45 mL/min
* Hepatic impairment with alanine aminotransferase or aspartate aminotransferase > 2 times the upper limit of normal, or Child-Pugh class B and C
* Malignant tumor within 3 years before Screening
* Memantine in any form, combination or dosage within 4 weeks prior to Screening
* Acetylcholinesterase inhibitors in any dosage form
* The subject has received active amyloid or tau immunization (i.e., vaccination for Alzheimer's disease) at any time, or passive immunization (i.e., monoclonal antibodies for Alzheimer's disease) within 6 months of Screening

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier San Martin, MD, Study Director — Chief Medical Officer
Locations (1):
- University of Rochester-AD-CARE Program, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Derived] Reda SM, Setti SE, Berthiaume AA, Wu W, Taylor RW, Johnston JL, Stein LR, Moebius HJ, Church KJ. Fosgonimeton attenuates amyloid-beta toxicity in preclinical models of Alzheimer's disease. Neurotherapeutics. 2024 Jul;21(4):e00350. doi: 10.1016/j.neurot.2024.e00350. Epub 2024 Apr 9. PMID 38599894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States.
Pre-assignment Details: This was a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the clinical efficacy of ATH-1017 treatment compared with placebo in participants with a clinical diagnosis of mild to moderate Alzheimer's disease (AD).
Groups:
- Placebo: Participants were randomized to receive placebo via subcutaneous (SC) injection once-daily (QD) preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- ATH-1017 40 Milligrams (mg): Participants were randomized to receive ATH-1017 40 mg via SC injection QD preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- ATH-1017 70 mg: Participants were randomized to receive ATH-1017 70 mg via SC injection QD preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
Period: Safety Population, >=1 Dose Administered
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg) | ATH-1017 70 mg
Started | 218 | 224 | 107
Completed | 183 | 174 | 69
Not Completed | 35 | 50 | 38
Not completed — Adverse Event | 10 | 22 | 18
Not completed — Withdrawal by Subject | 3 | 6 | 1
Not completed — Lost to Follow-up | 0 | 3 | 2
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Undetermined | 15 | 9 | 5
Not completed — >1 Reason | 4 | 7 | 12
Period: Primary Analysis Population
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg) | ATH-1017 70 mg
Started | 144 | 143 | 0
Completed | 128 | 122 | 0
Not Completed | 16 | 21 | 0
Not completed — Adverse Event | 6 | 9 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Undetermined | 7 | 3 | 0
Not completed — >1 Reason | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: included all randomized participants who received at least one dose of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg) | ATH-1017 70 mg | Total
Number analyzed (Participants) | 218 | 224 | 107 | 549
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (7.22) | 72.7 (7.24) | 71.0 (6.80) | 72.6 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 115 | 56 | 287
  Male | 102 | 109 | 51 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 45 | 6 | 90
  Not Hispanic or Latino | 179 | 177 | 101 | 457
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 7 | 1 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 14 | 19 | 8 | 41
  White | 185 | 194 | 97 | 476
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Global Statistical Test (GST) Score
Description: The Global Statistical Test (GST) score is a composite of cognition and function, calculated as the average of two change from baseline z-scores; the z-scores are calculated for the change from baseline scores for cognition (Alzheimer's Disease Assessment Scale-Cognitive Subscale [ADAS-Cog11]; lower value indicates improvement) and function (Alzheimer's Disease Cooperative Study - Activities of Daily Living, 23-item version [ADCS-ADL23] score; higher value indicates improvement).
  GST is a standardized score relative to the population mean. Therefore, a GST score of 0 is representative of the population mean. Since GST is a composite of two endpoints, a negative ADCS-ADL23 score is used in deriving GST. Therefore, a lower score indicates improvement, and a higher score indicates worsening. There are no defined clinically relevant thresholds for this GST score.
Time Frame: Baseline and Week 26
Population: Primary Analysis Population (Placebo or 40 mg ATH-1017 mITT Participants not taking AChEIs)
Measure: Least Squares Mean (Standard Error); unit: Z-score
Groups:
- ATH-1017 40 Milligrams (mg): Daily subcutaneous (SC) injection of 40mg ATH-1017
  ATH-1017: Daily subcutaneous (SC) injection of ATH-1017 in a pre-filled syringe
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg)
Number analyzed (Participants) | 144 | 143
Z-score | -0.126 (0.0683) | -0.208 (0.0707)

2. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog11) Change From Baseline
Description: The ADAS-Cog11 was designed to measure cognitive symptom change in participants with Alzheimer's Disease (AD) and consisted of 11 tasks. The standard 11 items (and corresponding score range) were: word recall (0-10), commands (0-5), constructional praxis (0-5), naming objects and fingers (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), spoken language ability (0-5), comprehension of spoken language (0-5), word-finding difficulty (0-5), and remembering test instructions (0-5). The test included 7 performance items and 4 clinician-rated items. The ADAS-Cog11 total score was the sum of all 11 individual items, with a total score ranging from 0 (no impairment) to 70 (severe impairment). Higher scores indicated more severe cognitive impairment. Baseline was defined as Day 1.
Time Frame: Baseline and Week 26
Population: Primary Analysis Population (Placebo or 40 mg ATH-1017 mITT Participants not taking AChEIs)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg)
Number analyzed (Participants) | 144 | 143
score on a scale | -0.39 (0.54) | -1.09 (0.56)

3. Secondary Outcome: Alzheimer's Disease Cooperative Study - Activities of Daily Living, 23-Item Version (ADCS-ADL23) Change From Baseline
Description: The ADCS-ADL23 is a 23-item assessment of functional impairment in terms of activities of daily living administered to the support person/caregiver. It comprises 23 questions about the subject's involvement and level of performance across items representing daily living. The questions range from basic to instrumental activities of daily living. Each item is rated from the highest level of independent performance to complete loss. The total score range is from 0 to 78, with lower scores indicating greater functional impairment. Baseline was defined as Day 1.
Time Frame: Baseline and Week 26
Population: Primary Analysis Population (Placebo or 40 mg ATH-1017 mITT Participants not taking AChEIs)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg)
Number analyzed (Participants) | 144 | 143
score on a scale | -0.02 (0.65) | 0.65 (0.67)

4. Secondary Outcome: Plasma Neurofilament Light Chain (NfL) Concentrations Change From Baseline
Description: Neurofilament light chain (NfL) is an objective biomarker of neurodegeneration and was measured to quantitatively support the evaluation of ATH-1017. Higher concentrations of NfL in plasma are associated with neurodegeneration.
Time Frame: Baseline and Week 26
Population: Primary Analysis Population (Placebo or 40 mg ATH-1017 mITT Participants not taking AChEIs)
Measure: Least Squares Mean (Standard Error); unit: picogram / milliter
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg)
Number analyzed (Participants) | 144 | 143
picogram / milliter | 2.95 (2.49) | -0.96 (2.48)

ADVERSE EVENTS:
Time Frame: Up to 30 weeks
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg) | ATH-1017 70 mg
All-Cause Mortality (participants affected / at risk) | 0/218 | 0/224 | 0/107
Serious Adverse Events (participants affected / at risk) | 15/218 | 11/224 | 3/107
Other Adverse Events (participants affected / at risk) | 65/218 | 185/224 | 104/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=218) | ATH-1017 40 Milligrams (mg) (N=224) | ATH-1017 70 mg (N=107)
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic arthropathy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=218) | ATH-1017 40 Milligrams (mg) (N=224) | ATH-1017 70 mg (N=107)
Injection site reactions (General disorders) | 31 | 128 | 78 — (high-level term)
COVID-19 (Infections and infestations) | 12 | 10 | 2
Urinary tract infection (Infections and infestations) | 9 | 5 | 2
Headache (Nervous system disorders) | 9 | 6 | 3
Fall (Injury, poisoning and procedural complications) | 9 | 10 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 10 | 6
Eosinophilia (Blood and lymphatic system disorders) | 0 | 16 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT04488419/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT04488419/SAP_001.pdf